CLINICAL TRIAL: NCT04629209
Title: A Phase II, Open Label Study of ONC201 in Adults With EGFR-low Glioblastoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in approach to study.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020LS093; ONC026 (Other: Chimerix)
Expanded Access: NCT04617002 (Approved for marketing)
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — TIC10 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: ONC201 with Surgical Resection in Glioblastoma (Experimental): Patients must be eligible for salvage surgical resection as deemed by the site Investigator. ONC201 will be administered orally, twice a week (2 consecutive days on and 5 days off per week) schedule at a dose of 625mg.
  Interventions: Drug: ONC201
- Arm B: ONC201 in Glioblastoma (Experimental): Unequivocal evidence of recurrence (progressive disease) on contrast-enhanced brain CT or MRI as defined by RANO criteria, or have documented recurrent glioma on diagnostic biopsy. ONC201 will be administered orally, twice a week (2 consecutive days on and 5 days off per week) schedule at a dose of 625mg.
  Interventions: Drug: ONC201

INTERVENTIONS:
Drug: ONC201 — ONC201 is a orally active, small molecule DRD2 antagonist that kills cancer cells but not normal cells.

SUMMARY:
This is an open-label, two arm study. The trial will enroll a total of up to 36 patients. Arm A will enroll up to a total of 6 evaluable patients and Arm B will enroll up to a total of 30 evaluable patients. Arm A will explore the intra-tumoral ONC201 concentrations and pharmacodynamic activity in adult EGFR-low glioblastoma patients. Arm B will determine the radiographic efficacy of ONC201 in adult recurrent EGFR-low glioblastoma patients. All patients will be treated with oral ONC201 (625 mg) twice weekly, 2 consecutive days on and 5 days off per week schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologically confirmed World Health Organization Grade IV glioblastoma.
2. Patient must have all of the following in their most recently resected archival tumor tissue: (1) absence of EGFR gene amplification by FISH, (2) absence of EGFRvIII expression by RT-PCR, and (3) low EGFR expression by IHC.
3. For Arm A: Patients must be eligible for salvage surgical resection as deemed by the site Investigator.

   For Arm B: Unequivocal evidence of recurrence (progressive disease) on contrast-enhanced brain CT or MRI as defined by RANO criteria, or have documented recurrent glioma on diagnostic biopsy.
4. Patient must have measurable disease by RANO criteria.
5. Patient must have had previous therapy with at least radiotherapy.
6. Patient must have an interval of at least 90 days from the completion of radiotherapy prior to the first dose of ONC201. If patients are within 90 days of radiotherapy, they may still be eligible if they meet one or more of the following criteria.

   * Progressive tumor is outside the original high-dose radiotherapy target volume as determined by the treating investigator, or
   * Histologic confirmation of tumor through biopsy or resection, or Nuclear medicine imaging, MR spectroscopy, or MR perfusion imaging consistent with true progressive disease, rather than pseudoprogression or radiation necrosis, obtained within 28 days of registration.
7. From the projected start of ONC201, the following time periods must have elapsed: 5 half-lives from any investigational agent, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from antibodies, or 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies.
8. All adverse events Grade > 1 related to prior therapies (chemotherapy, radiotherapy, and/or surgery) must be resolved to grade 1 or baseline, except for alopecia and sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment, are acceptable.
9. Patient must be ≥18 years of age.
10. Patient must have a Karnofsky Performance Status (KPS) ≥ 60
11. Patient must have adequate organ and marrow function as defined below, all screening labs should be performed within 14 days of treatment initiation:

    * leukocytes ≥ 3,000/mcL
    * absolute neutrophil count ≥ 1,500/mcL
    * platelets ≥ 75,000/mcL
    * hemoglobin > 8.0 mg/dL
    * total bilirubin ≤ 2.0 x upper limit of normal
    * AST (SGOT)/ALT (SGPT) ≤ 2.5 × upper limit of normal
    * creatinine ≤ ULN OR creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above normal.
12. Patient must have a contrast-enhanced head CT or brain MRI and total spine MRI within 14 days prior to start of study drug.
13. Corticosteroid dose must be stable or decreasing for at least 3 days prior to the baseline CT or MRI scan.
14. The effects of ONC201 on the developing human fetus are unknown. For this reason, women of childbearing potential (WOCBP) and men must agree to use adequate contraception prior to study entry and for the duration of study participation and for 30 days after the last dose of therapy. Highly effective contraceptive measures include: stable use of oral contraceptives such as combined estrogen and progestogen and progestogen only hormonal contraception or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; intrauterine hormone- releasing system (IUS); bilateral tubal ligation; vasectomy and sexual abstinence.
15. WOCBP must have a negative serum or urine pregnancy test within 28 days of initiation of dosing.
16. Contraception is not required for men with documented vasectomy.
17. Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of childbearing potential.
18. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.
19. Availability of formalin-fixed paraffin-embedded tumor tissue.
20. Patient must have the ability to be able to swallow and retain orally administered medication.
21. Patient must have the ability to understand and the willingness to sign a written informed consent document. Only patients who have capacity to consent will be enrolled in the study.

Exclusion Criteria:

1. Patient has a midline glioma.
2. Patient has a known histone H3 K27M mutation.
3. Patient has a known IDH1 (isocitrate dehydrogenase 1) or IDH2 mutations or 1p/19q co-deletion.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ONC201 or its excipients (See Section 8).
5. Presence of diffuse leptomeningeal disease or evidence of CSF dissemination.
6. Current or planned participation in a study of an investigational agent or using an investigational device.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
8. Active infection requiring systemic therapy.
9. Pregnant and/or breastfeeding women or unable to maintain use of contraception while on study and for 30 days after the last dose of study drug.
10. Known HIV-positive test on combination antiretroviral therapy.
11. Known history of cardiac arrhythmias including atrial fibrillation, tachyarrhythmias or bradycardia, unless arrhythmia is controlled and after Cardiology has cleared patient to receive ONC201.
12. History of CHF, or MI or stroke in the last 3 months.
13. Receiving therapeutic agents known to prolong QT interval.
14. Active illicit drug use or diagnosis of alcoholism that would interfere with study compliance or the assessment of outcomes.
15. Known additional malignancy that is progressing or requires active treatment within 3 years of start of study drug. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ melanoma, or in situ cervical cancer that has undergone potentially curative therapy.
16. Any surgery (not including minor diagnostic procedures such as lymph node biopsy) within 2 weeks of baseline disease assessments; or not fully recovered from any side effects of previous procedures. An interval of 1 week for stereotactic brain biopsy from the start of ONC201 is acceptable.
17. Concomitant use of potent CYP3A4/5 inhibitors during the treatment phase of the study and within 72 hours prior to starting ONC201.
18. Concomitant use of potent CYP3A4/5 inducers, which include enzyme inducing antiepileptic drugs (EIAEDs) (see Appendix B), during the treatment phase of the study and within 2 weeks prior to starting ONC201. Concurrent dexamethasone is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-28 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Intra-tumoral ONC201 concentrations | 11 Days
  intra-tumoral ONC201 concentrations in adult EGFR-low glioblastoma patients. The drug concentrations will be measured in micrograms per milliliters.
Objective Response Rate | 6 months
  Objective Response Rate of ONC201 in adult recurrent EGFR-low glioblastoma patients. Measured using the RANO criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No